CLINICAL TRIAL: NCT04918732
Title: Identification and Characterization of Non-alcoholic Fatty Liver Disease in Primary Care
Brief Title: NAFLD Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METC20-051
Record Dates: First submitted 2021-05-19; First posted 2021-06-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Cardiovascular Diseases; Type2 Diabetes; Metabolic Syndrome; Overweight and Obesity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Cardiovascular Diseases; Metabolic Syndrome; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FibroScan — The FibroScan device developed by Echosens (France) measures the liver stifness and steatosis based on a pulse of sound waves that goes through the liver.

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is with 25% the most prevalent liver disorder in Western society and is associated with overweight, obesity, metabolic syndrome (MetS), type 2 diabetes mellitus (T2DM), cardiovascular diseases (CVD) and increased risk of cancer development. NAFLD is defined by a hepatic fat accumulation of more than 5% in the absence of classical causes of steatogenesis (e.g. alcohol and steatogenic drugs). It represents a broad spectrum of clinical entities from non-alcoholic fatty liver (NAFL) to advanced liver disease with hepatic failure. Most of the patients have simple steatosis, however in about 15-30% non-alcoholic steatohepatitis (NASH) develops, which leads to an overall increase in morbidity and mortality due to the progression to fibrosis, cirrhosis and hepatocellular carcinoma (HCC). Patients with NAFLD have no or few, mainly aspecific symptoms; and generally there is a silent progression of simple steatosis to NASH and in the end liver-related morbidity and mortality. Despite the clinical importance and the potential impact on healthcare resources, there is a striking lack of awareness on all levels of NAFLD. Furthermore, little to know data are available concerning the quality of life of NAFLD patients. Additionally, the majority of NAFLD patients are currently not detected due to the lack of non-invasive methods to diagnose NAFLD. Most of these patients, as a first contact in the healthcare system, will be found in the outpatient clinic of the general practitioner (GP). To date, it is not clear what the burden is of NAFLD and related diseases in at risk subjects in primary care. Therefore, identification of NAFLD patients in this cohort will give information on the prevalence in the group of uncomplicated overweight and obesity and those with concomitant cardiometabolic diseases. By early detecting these patients at risk to develop progressive liver diseases and extrahepatic manifestations, it will be possible to intervene and improve health.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign the informed consent
* Able to speak Dutch
* Between 18-80 years
* BMI >25 kg/m²
* Having one of the following conditions: 1)overweight, 2) obesity, 3) type 2 diabetes mellitus, 4) cardiovascular diseases (hypertension, atherosclerosis, angina pectoris, ischaemic heart condition, cerebrovascular condition)

Exclusion Criteria:

* Excessive alcohol use (more than 20 g/day for women and 30g/day for men= >2 glasses alcohol/day for women and >3 glasses for men)
* Other liver diseases: Hepatitis B virus, Hepatitis C virus, autoimmune hepatitis, primary biliary cirrhosis, hemochromatosis, Wilson's disease, Alpha 1 antitrypsin deficiency
* Secondary causes for steatosis: disorders of lipid metabolism, HCV Genotype 3, total parental nutrition, severe surgical weight loss, medications (amiodarone, tamoxifen, methotrexate, corticosteroids and HAART), lean steatosis, Celiac disease, environmental toxicity
* Pregnancy and breastfeeding.
* A history of bariatric surgery.
* Diagnosis of liver cirrhosis and/or hepatocellular carcinoma.
* Current diagnosis of extrahepatic malignancy(s) or prior diagnosis within last 5 years.
* Individuals about to undergo a surgery or otherwise medical procedure that will interfere with data collection and analyses planned within the current cohort, will initially be excluded from participation, but are offered the opportunity to participate at a later moment in time (e.g., after 3 months are myocardial infarction patients are eligible for participation).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1470 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of NAFLD in risk groups followed by the general practitioner | 3 years

SECONDARY OUTCOMES:
To study the risk factor overweight in the development of NAFLD | 3 years
  To see if there is an effect of having a BMI between 25 and 30 kg/m² in the development of NAFLD. The physiological parameter used will be BMI.
To study the risk factor obesity in the development of NAFLD | 3 years
  To see if there is an effect of having a BMI between 30-40 kg/m² on the development of NAFLD. The physiological parameter used will be BMI.
To study the risk factor metabolic syndrome in the development of NAFLD | 3 years
  To see if there is an effect of metabolic syndrome (defined by the criteria of the International Diabetes Federation) on the development of NAFLD.
To study the risk factor type 2 diabetes mellitus in the development of NAFLD | 3 years
  Type 2 diabetes mellitus will be assessed based on previous diagnosis and HbA1c levels.
To study the risk factor cardiovascular diseases in the development of NAFLD | 3 years
  Cardiovascular diseases will be assessed based on medical history found in the EPF.
To assess if the patient has a depression | 3 years
  Depression will be assessed using the patient-health questionnaire 9 (PHQ-9).
To assess if the patient has a anxiety issues | 3 years
  Anxiety will be assessed using the general anxiety disorder questionnaire (GAD-7)
To assess if the general wellbeing of the patient. | 3 years
  General wellbeing will be assessed using the short-health form-36 (SF-36).
To assess the physical state of the patient. | 3 years
  The physical state will be assessed using the BAECKE questionnaire.
To assess the work productivity and absenteism of the patient. | 3 years
  The work productivity will be assessed using the WPAI-SHP questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands